CLINICAL TRIAL: NCT03011697
Title: A Prospective, Single-center,Registry Study of Chinese Hospitalized Adult Patients With Valvular Heart Disease
Brief Title: Valvular Heart Disease Registry Study in Second Affiliated Hospital of ZheJiang University
Acronym: VHD-ZJU
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Jian'an Wang,MD,PhD, President of Second Affiliated Hospital, School of Medicine, Zhejiang University & Chief of Cardiology, Second Affiliated Hospital, School of Medicine, Zhejiang University
Other Study IDs: SAHZJU CT010
Record Dates: First submitted 2017-01-04; First posted 2017-01-05 (Estimated); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Valvular Heart Disease
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
We design a prospective, observational cohort study to provide contemporary information on the prevalence, characteristics, risk stratification，cost-effective ,treatments and prognosis of Chinese hospitalised adult patients with valvular heart disease.

DETAILED DESCRIPTION:
Valvular heart disease (VHD) is becoming more and more frequent with the aging, which has brought a heavy burden to the world. However, the prevalence and prognosis of valvular heart disease are not so clear, especially in the developing countries such as China etc. Because of the slow and progressive nature of VHD, symptoms might not be too severe to be diagnosed on time. Our retrospective survey (Int J Cardiol. 2016 Nov 25) indicated that severe valvular diseases are very common in China. Hence, we design a prospective, observational cohort study to provide contemporary information on the prevalence, characteristics, risk stratification，cost-effective ,treatments and prognosis of Chinese hospitalised adult patients with valvular heart disease.

ELIGIBILITY:
Inclusion Criteria:

Hospitalized patients over 18 years old meet one of the following conditions.

1. moderate or above valvular heart disease as defined by echocardiography: 1.1 Aortic stenosis, moderate or above, or valve area ≤1.5cm2, or maximal jet velocity ≥3.0m/sec, or mean pressure gradient ≥20mmHg, 1.2 Aortic regurgitation, moderate or above, or jet width ≥25% of left ventricular outflow tract, or regurgitant volume ≥30ml/beat, or regurgitant fraction ≥30%, 1.3 Mitral stenosis, moderate or above, or valve area ≤2.0cm2, 1.4 Mitral regurgitation, moderate or above, or effective regurgitant orifice ≥0.2cm2, or regurgitant volume ≥30ml/beat, or regurgitant fraction ≥30%, 1.5 Tricuspid stenosis, moderate or above, or valve area ≤1.0cm2, 1.6 Tricuspid regurgitation, moderate or above, or central jet area ≥5.0cm2, 1.7 Pulmonic stenosis, moderate or above, or maximal jet velocity >4m/sec, 1.8 Pulmonic regurgitation, moderate or above,
2. Patients who had undergone any operation on a cardiac valve (percutaneous balloon commissurotomy, valve repair, valve replacement, transcatheter aortic valve implantation),
3. Diagnosis of endocarditis as assessed by Duke criteria.

Exclusion Criteria:

1. Patients cannot be followed up for any reasons.
2. Patients in critical condition may be die in one year.
3. Patients have been enrolled in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 10000 hospitalized patients over 18 years old with valvular heart disease will be enrolled consecutively
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality and disabling strokes | one year
  All-cause mortality and disabling strokes

SECONDARY OUTCOMES:
Hospitalization for heart failure | one year
  Hospitalization for heart failure
Surgical or transcatheter aortic valve replacement | one year
  Surgical or transcatheter aortic valve replacement

CONTACTS AND LOCATIONS:
Overall Officials: Wang Jian-an, MD,PhD, Principal Investigator — Second Affiliated Hospital Zhejiang University School of Medicine
Locations (1):
- 2nd Affiliated Hospital, School of Medicine at Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Hu P, Liu XB, Liang J, Zhu QF, Pu CX, Tang MY, Wang JA. A hospital-based survey of patients with severe valvular heart disease in China. Int J Cardiol. 2017 Mar 15;231:244-247. doi: 10.1016/j.ijcard.2016.11.301. Epub 2016 Nov 25. PMID 27908608
- See also: hospital-based survey of patients with severe valvular heart disease in China — http://www.ncbi.nlm.nih.gov/pubmed/27908608